CLINICAL TRIAL: NCT06966791
Title: Examınatıon of Sexual Functıon in Young Women After Breast Cancer Surgery
Brief Title: Sexual Functıon in Young Women After Breast Cancer Surgery
Status: Recruiting | Type: Observational
Sponsor: ATİYE KAŞ ÖZDEMİR (Other)
Responsible Party: Sponsor-Investigator, ATİYE KAŞ ÖZDEMİR, Principal Investigator, Pamukkale University
Organization: Pamukkale University (Other)
Other Study IDs: E-60116787-020-631173
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Surgery; Young Adult Females
Keywords: sexual functions; breast cancer surgery; young adult females; Breast Cancer Treatment; quality of life; breast cancer survival; body perception; Mastectomy; Mastectomy, Modified Radical; Mastectomy, Segmental; breast conserving surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young women with breast cancer: Sexually active young women scheduled for breast cancer surgery
  Interventions: Other: No intervention will be performed as part of this study. However, regardless of the study, all participants will have breast cancer surgery

INTERVENTIONS:
Other: No intervention will be performed as part of this study. However, regardless of the study, all participants will have breast cancer surgery — No intervention will be performed as part of this study. However, regardless of the study, all participants will have breast cancer surgery and other breast cancer treatments.

SUMMARY:
The aim of this observational study was to analyse sexual function in young women after breast cancer surgery. The main question it aims to answer is Sexual function in young women after breast cancer surgery changes during the one-year follow-up period. Participants will answer demographic information, Female Sexual Function Scale, Breast-Q and Body Perception Scale about their sexual function, quality of life and body perception. These will be recorded before surgery and repeated 6 weeks, 6 months and 1 year after surgery.

DETAILED DESCRIPTION:
As a result of the power analysis of the preliminary study conducted with the participation of 9 cases; it was calculated that 80% power could be obtained at 95% confidence level when at least 47 people were included in the study. However, considering that the results of the preliminary study will not be conclusive, it is planned to complete the study with at least 52 people by taking 10% more participants. The data will be analysed with SPSS 25.0 package programme. Continuous variables will be given as mean ± standard deviation and categorical variables as number and percentage. Repeated measures ANOVA test, Kruskal-Wallis test or Friedman test will be used according to the parametric test assumptions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals scheduled for surgery for breast cancer
* Accepting to participate in the study
* Being sexually active in the last 1 year
* Continuation of menstruation

Exclusion Criteria:

* Previous breast cancer surgery
* Previous history of breast cancer
* History of any other cancer
* Refusal to participate in the study
* Refusal to continue working
* Problems in her relationship with her partner

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Study Population: Individuals who are followed up by Pamukkale University Breast Polyclinic
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sexual function | It is planned to repeat the measurements 4 times: before, 6 weeks, 6 months and 12 months after breast cancer surgery.
  In this study, it is planned to follow up the patients from the early postoperative period in order to emphasise and draw attention to the difficulties experienced by individuals with breast cancer in their sexual life. Female sexual function will evaluate with a detailed 19-item likert-type questionnaire [Female Sexual Function Index (FSFI)] described by Rosen et al.
  Questions 1 and 2 are scored between 1-5, questions 3-13 are scored between 0-5, questions 14-16 are scored between 0 and 1-5 and questions 17-19 are scored between 0-5. Accordingly, the highest raw score to be obtained from the scale is 95 and the lowest raw score is 4. The cut-off score of the scale is determined as 26.55 and it is stated that women who score below this score have sexual dysfunction (Aydemir and Güneş 2024). High scores on the scale indicate that sexual function is good. The Turkish validity and reliability study of the scale was conducted by Aygin and Aslan in 2005.

SECONDARY OUTCOMES:
Quality of life of participants | It is planned to repeat the measurements 4 times: before, 6 weeks, 6 months and 12 months after breast cancer surgery.
  Breast-Q, a validated, patient-reported outcome measure, will be used to assess the satisfaction and quality of life of patients undergoing breast cancer surgery.The breast satisfaction section consists of 4 questions scored 1-4, the psychosocial well-being section consists of 10 questions scored 1-5, the sexual well-being section consists of 6 questions scored 1-5, the physical well-being section consists of 10/11 questions scored 1-3, and the radiation side effects section consists of 6 questions scored 1-3. Higher scores represent better results.
Participants' body perception | It is planned to repeat the measurements 4 times: before, 6 weeks, 6 months and 12 months after breast cancer surgery.
  The Body Perception Scale developed by Secord and Jourand will be used to evaluate the body perception of the participants.The scale consists of 40 items, each item related to an organ or a part or function of the body. The scale, which offers a Likert-type scoring between 1-5 for each item as 'I don't like it at all', 'I don't like it', 'I don't like it', 'I am undecided', 'I like it' and 'I like it very much', is scored between 40-200 in total. The cut-off score of the scale is 135, and those with a score below 135 are defined as the group with low body image (Hamurcu et al. 2015).

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No